CLINICAL TRIAL: NCT02608762
Title: Neurobehavioral Outcomes and Quality of Life in Pediatric Patients With Brain or Head/Neck Tumors Receiving Proton or Photon Radiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-5729A3
Record Dates: First submitted 2015-10-29; First posted 2015-11-20 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Brain Tumor
Keywords: Pediatric brain tumors; Radiation therapy; Neurobehavioral functions; Proton radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pediatric/adolescent patients with brain tumors: A prospectively recruited of newly-diagnosed pediatric/adolescent patients with brain tumors or head/neck cancers
  Interventions: Radiation: standard adjuvant local radiation therapy or cranial radiation therapy

INTERVENTIONS:
Radiation: standard adjuvant local radiation therapy or cranial radiation therapy

SUMMARY:
Background: Neurobehavioral functions and quality of life (QoL) are the important outcome measurements after radiotherapy in patients with brain tumors and even head/neck cancers. However, few studies have focused on neurobehavioral functions and QoL after anti-cancer treatment particularly brain radiotherapy for pediatric/adolescent patients with brain tumors. This study thus aims to prospectively evaluate those functions in pediatric or adolescent patients with brain or head/neck tumors in order to provide useful information about their clinical outcomes.

Methods: A total of 72 pediatric/adolescent patients, who are diagnosed with brain tumors or head/neck cancers, were prospectively recruited. Neurobehavioral functions will be evaluated using a neuropsychological battery, which includes general cognitive functions, intelligence, memory, executive functions, information processing and emotional/behavioral expressions. The QoL will be evaluated by the health-related QoL questionnaire. All participants will be examined at six phases, which include pre-treatment, 1-month post-treatment, 4-month post-treatment, 1-year post-treatment, 2-year post-treatment and 3-year post-treatment.

Expected results: Patients'neurobehavioral functions and QoL will show significant improvement after treatment, and the improvement will not be diminished across each post-treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with brain tumors or head/neck cancers who are no older than 18 years old
* Patients should be considered indicated for receiving the subsequent course of local radiotherapy

Exclusion Criteria:

* Patients who received radiotherapy once before
* Patients have visual and/or hearing impairments which obviously impede the administration of neurocognitive assessment
* Patients cannot underwent brain MRI examination because of clinical contraindications, such as renal insufficiency (GFR <30)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric/adolescent patients, who are diagnosed with brain tumors or head/neck cancers, were prospectively recruited.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in Intellectual functioning from baseline to 3 months after the start of radiotherapy | 1 week before the start of radiotherapy and 3 months after the start of radiotherapy
  Intellectual functioning mainly includes subtests of Wechsler Intelligence scale for Children
Neurobehavioral functions and psychosocial adjustments | 3 months after the start of radiotherapy
  In this study, evaluations of neurocognitive functions include memory scores of verbal memory (NEPSY-II),memory scores of non-verbal memory (NEPSY-II) raw scores of executive functions (NEPSY-II), raw scores of processing speed (NEPSY-II), raw scores of attention (Continuous Performance Test, CPT).
  Evaluations of psychosocial adjustments mainly include severity scores of behavioral problems (Achenbach System of Empirically Based Assessment),scores of behavioral problems(Vineland Adaptive Behavior Scale), scores of parental stress (Parenting Stress Index, PSI) and scores on the scale for quality of life (Child Health Questionnaire, CHQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan